CLINICAL TRIAL: NCT07256665
Title: The Cracking Consciousness Study With Monroe & Neuphoria
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Efforia, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 41035
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Mental Energy; Stress

STUDY DESIGN:
Intervention Model Description: Single Arm observational where participants act as their own control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm longitudinal where participants act as their own control (Experimental): Single Arm longitudinal where participants act as their own control
  Interventions: Device: Neuphoria Wearable

INTERVENTIONS:
Device: Neuphoria Wearable — Neuphoria wearable measures Electroencephalography (EEG) brainwaves.

SUMMARY:
You've explored the Monroe Focus levels. But, Bob Monroe said, "You might believe something, but you won't understand it until you can measure it with objective data." Now, for the first time, we can measure them. In partnership with Neuphoria, we're launching a groundbreaking EEG study to define Higher States of Consciousness. Join the World's First higher states of Consciousness Study.

DETAILED DESCRIPTION:
This remotely administered decentralized trial is designed to explore the potential of the Neuphoria device, a cutting-edge wearable neurofeedback headset, in enhancing cognitive performance and facilitating the attainment of peak mental states. By leveraging advanced EEG technology to monitor brainwave activity in real-time, this study aims to provide participants with personalized feedback, assisting them in training their brains to improve focus, creativity, and achieve flow states. The device serves as a comprehensive brain optimization platform, offering personalized assessments, data-driven insights, and actionable recommendations for mental well-being.

In an era where mindfulness and meditation are highly valued, yet often unquantified, this study emerges as a pioneering effort to measure these elusive higher states of consciousness scientifically. In collaboration with Neuphoria, this trial endeavors to blend the art of introspection with the precision of EEG technology, thereby transforming belief into understanding and folklore into facts. The ultimate goal is to redefine mental wellness by gaining a deeper understanding of consciousness shifts.

Participants in this trial are invited to embark on a unique journey of self-discovery, exploring their mental landscapes while capturing data that reflects their progress toward higher consciousness. Through engagement with meditation and mindfulness techniques, participants will not only gain insights into their stress levels and mindfulness tendencies, quantified through tools like the Perceived Stress Scale and the Freiburg Mindfulness Inventory, but also discover their personal pathways to enhanced mental wellness and consciousness.

The study's primary aim is to objectively measure shifts in participants' consciousness using EEG data, in conjunction with traditional mindfulness and stress metrics. By offering personalized insights into the effects of meditation and mindfulness on mental health, the study empowers participants to make informed decisions regarding their self-care practices.

The significance of this trial lies in its potential to transform subjective meditation experiences into objective, measurable data, thereby narrowing the gap between belief and measurable outcomes. Understanding the influence of mindfulness practices on consciousness could significantly advance mental health optimization strategies. While acknowledging the limitations in the universal applicability of its results, the personalized insights provided by this study promise to be invaluable for participants eager to deepen their mindfulness practice and achieve a state of equanimity. Through this innovative, remotely administered trial, we aim to illuminate the path to mental wellness and elevated consciousness for individuals across the globe.

ELIGIBILITY:
Inclusion Criteria:

* Can read and understand English.
* US resident.
* Willing and able to follow the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-10 (Actual); Primary Completion 2026-08-10 (Estimated); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
Neuphoria Brain EEG | Change from baseline (Day 1-7) in cognitive and physiological profiles at 4 to 5 weeks (Day 23-37) after the start of the intervention
  Neuphoria's wearable neurofeedback system harnesses real-time EEG to generate a rich, multidimensional cognitive profile by measuring five core metrics-mental state, mindset, nervous system activity, emotion, and breathing patterns-all displayed via its biohacking dashboard to offer users nuanced insights into their cognitive and physiological functioning
Perceived Stress Scale (Past Week Version) | Change from baseline (Day 1-3) in perceived stress levels at 4 to 5 weeks (Day 27-33) after the start of the intervention
  The Perceived Stress Scale (Past Week Version) is a modified version of the classic stress assessment tool that evaluates stress levels based on recent experiences within the last week. This scale helps in understanding how various situations have recently affected an individual's feelings and perceived stress levels. By focusing on a shorter time frame, it provides a more immediate assessment of stress, which can be particularly useful for quickly evaluating the effectiveness of stress management strategies or interventions. The tool retains its original structure, ensuring its reliability while making it more relevant for current stress evaluation.
Freiburg Mindfulness Inventory | Change from baseline (Day 1-3) in mindfulness levels at 4 to 5 weeks (Day 27-33) after the start of the intervention
  The Freiburg Mindfulness Inventory (FMI) is a valid and reliable questionnaire designed to measure mindfulness. The 14 items in the inventory cover all aspects of mindfulness. Participants are asked to reflect on their experiences over a certain period of time and answer each statement as honestly and spontaneously as possible. There are no 'right' or 'wrong' answers, the focus is solely on personal experience.

CONTACTS AND LOCATIONS:
Locations (1):
- Efforia, New York, New York, United States

REFERENCES:
- See also: Additional information and join instructions on Efforia — https://app.efforia.com/wp-admin/admin.php?page=llms-course-builder&course_id=41035